CLINICAL TRIAL: NCT05268224
Title: Investigation of a Tear-based, Lab-developed Biological Test for Breast Cancer, as a Supplemental Tool to Current Screening Recommendations for Women With Dense Breast Tissue.
Brief Title: A Tear-based, Lab-developed Test for Breast Cancer for Women With Dense Breast Tissue
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Namida Lab (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB#2022-0073
Record Dates: First submitted 2022-02-24; First posted 2022-03-07 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dense Breast: Women mammographically categorized as having either heterogeneously dense or extremely dense breast tissue.
  Interventions: Diagnostic Test: Schirmer Strip

INTERVENTIONS:
Diagnostic Test: Schirmer Strip — A tear-based screening assay for breast cancer developed and validated by Namida Lab, Inc., a high complexity CLIA-certified lab. It consists of two parts: tear sample collection using a Schirmer Strip and a clinical lab-developed test that measures protein biomarkers for breast cancer screening.

SUMMARY:
Investigation of a tear-based, lab-developed biological test for breast cancer, as a supplemental tool to current screening recommendations for women with dense breast tissue will explore if a tear-based biological test can be used as a support tool in the breast cancer screening protocol for women with dense breast tissue. The test was designed and validated by Namida Lab, Inc., a high complexity Clinical Laboratory Improvement Amendments (CLIA) certified lab.

ELIGIBILITY:
Inclusion Criteria:

Categorized as having heterogeneously dense or extremely dense tissue 18 years of age or older Able to understand the informed consent process Willing to comply with all study procedures

Exclusion Criteria:

Have an active eye infection Categorized as having fibro glandular densities or fatty breast tissue Currently diagnosed or are receiving treatment for breast cancer Under 18 years of age

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is based on individuals who biologically qualify to participate in yearly breast cancer screening and who have dense breast tissue.
Study Population: Women who have been mammographically catagorized as having heterogenously dense or extremely dense breast tissue.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Accuracy Measure | 3 months
  Degree of closeness of categorization by a tear-based biological test scores to imaging techniques

CONTACTS AND LOCATIONS:
Locations (1):
- Namida Lab, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not intended to be shared with other researchers at this time.